CLINICAL TRIAL: NCT00994734
Title: Uptake and Acceptability of Home-use of Mifepristone for Medical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1.2.3
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Termination of Pregnancy
MeSH Terms: interventions — Mifepristone

ARMS (2):
- clinic administration of mifepristone (No Intervention)
- home administration of mifepristone (Experimental)
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — home administration of mifepristone
  Arms: home administration of mifepristone

SUMMARY:
The primary aim of this study is to assess the acceptability of home-use mifepristone for termination of pregnancy among women who choose it and their providers. The investigators' secondary aims are to assess rates of follow-up, adherence, efficacy, complications, lost productivity, and to estimate the minimum proportion of women who choose home-use over clinic use of mifepristone.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age women seeking abortion services.
* Eligible women will be in general good health and assessed by a clinician to have an intrauterine pregnancy less than 64 days L.M.P on the day mifepristone will be taken.
* Participants must be eligible for medical abortion according to clinician and clinic standards.
* In the United States, women only 18 years and older will be eligible to participate, unless the study site obtains a waiver to include minors.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 615 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Proportion of women who select home-use of mifepristone | 1-2 weeks
Satisfaction with Method | 1-2 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Feminist Women's Health Center, Atlanta, Georgia
  - Institute for Family Health, New York, New York
  - Family Health Center, Montefiore Medical Center, The Bronx, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Municipal Clinical Hospital, Chisinau, Moldova
- Nepal (2):
  - Kathmandu Medical College, Kathmandu
  - Nepal Medical College Teaching Hospital, Kathmandu

REFERENCES:
- [Derived] Conkling K, Karki C, Tuladhar H, Bracken H, Winikoff B. A prospective open-label study of home use of mifepristone for medical abortion in Nepal. Int J Gynaecol Obstet. 2015 Mar;128(3):220-3. doi: 10.1016/j.ijgo.2014.09.022. Epub 2014 Nov 27. PMID 25482435